CLINICAL TRIAL: NCT05344144
Title: The Effect of Emotional Freedom Technique and Music, Applied to Pregnant Women Having Experienced Prenatal Loss on Psychological Development, Well-Being Status and Cortisol Levels
Brief Title: EFT and Music on Psychological Development, Well-Being Status and Cortisol Level in Pregnant Women
Acronym: EFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Esra KARATAŞ OKYAY, Principal Investigator, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KSUESRAKARATASOKYAY001
Record Dates: First submitted 2022-04-01; First posted 2022-04-25 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Pregnancy Loss; Anxiety
Keywords: Emotional Freedom Technique; Midwifery; Well-Being Status; Cortisol; Music; Prenatal loss; Psychological Development
MeSH Terms: conditions — Anxiety Disorders | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Emotional freedom technique group (Experimental): Emotional freedom technique group pregnant women who have experienced prenatal loss, who were included in the emotional freedom technique group with randomization method, will be given a counseling program including psychosocial care and emotional freedom technique application in addition to the routine.
  Interventions: Other: Emotional Freedom Technique
- Music group (Experimental): Music group pregnant women who have experienced prenatal loss, who were included in the music group with randomization method, will be given a counseling program including music application in addition to the routine.
  Interventions: Other: Music
- Control (No Intervention): control group standard care group

INTERVENTIONS:
Other: Emotional Freedom Technique — EFT was applied to pregnant women with a history of prenatal loss twice, one week apart, by the researcher. Between the two treatments, they were given personalized homework (on waking up in the morning and before going to sleep at night) for self-administration.
  Arms: Emotional freedom technique group
Other: Music — Music practice was applied to the pregnant women with a history of prenatal loss twice, one week apart, by the researcher. For one week after the first application, the music application was applied by the pregnant woman once a day/for 30 minutes, and the researcher was reminded by phone message.
  Arms: Music group

SUMMARY:
Emotional freedom technique and music were applied to pregnant women who experienced prenatal loss. Emotional freedom technique group, music group and control groups each consisted of 53 pregnant women.

DETAILED DESCRIPTION:
Aim: The research is conducted to determine for the purpose of the effect of emotional freedom technique and music applied to pregnant women having experienced prenatal loss on psychological development, well-being status, and cortisol level.

Material and Method: The research is conducted in a randomized controlled manner with a total of 159 pregnant women who applied to the gynecology outpatient clinics of Elazig Fethi Sekin City Hospital between October 2020 and April 2021 (53 EFT, 53 music, 53 control). In the research, EFT was applied to the pregnant women in the EFT group twice, with an interval of one week; pregnant women in the music group were listened to music twice, with a one-week interval. Pregnant women continued the attempts for one week after the first attempt. SUDS, SUE Scale, PTGI, WHO-5 WellBeing Index were used to collect data, and a saliva sample was taken.

ELIGIBILITY:
Inclusion Criteria:

1. Anxiety level is 1 and above when measured with the subjective discomfort unit scale (Appendix 3),
2. 18 years old and over,
3. There are no conditions such as infection, wound, scar in the tapping areas,
4. All pregnant women who did not have any health problems (such as preeclampsia, diabetes, heart disease, placenta previa, oligohydramnios, fetal anomaly) during pregnancy and baby were included in the sample.

Exclusion Criteria:

1. Having any problem that prevents communication (such as not knowing Turkish, having hearing, speaking and understanding abilities),
2. Contaminated salivary cortisol,
3. Those with psychiatric health problems according to their medical records were excluded from the study.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 159 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-10-06 (Actual)

PRIMARY OUTCOMES:
Determining the level of anxiety | In the first interview, SUE was applied to all pregnant women in all three groups as a pre-test at any time of pregnancy.
  In order to determine the anxiety level of the pregnant women, SUE (Subjective Units of Experience) was applied. SUE is used to determine the intensity of the person's emotion at the beginning and end of therapy. The scale is scored between -10 and +10, with negative numbers for negative/unpleasant experiences and positive numbers for positive/pleasant experiences.
Determining the level of anxiety | One hour after the first interview, SUE was applied to all pregnant women in all three groups.
  In order to determine the anxiety level of the pregnant women, SUE was applied. SUE is used to determine the intensity of the person's emotion at the beginning and end of therapy. The scale is scored between -10 and +10, with negative numbers for negative/unpleasant experiences and positive numbers for positive/pleasant experiences.
Determining the level of anxiety | Seven day after the first interview, SUE was applied to all pregnant women in all three groups.
  In order to determine the anxiety level of the pregnant women, SUE was applied. SUE is used to determine the intensity of the person's emotion at the beginning and end of therapy. The scale is scored between -10 and +10, with negative numbers for negative/unpleasant experiences and positive numbers for positive/pleasant experiences.
Determining the level of anxiety | One hour after the third measurement, SUE was applied to all pregnant women in all three groups.
  In order to determine the anxiety level of the pregnant women, SUE was applied. SUE is used to determine the intensity of the person's emotion at the beginning and end of therapy. The scale is scored between -10 and +10, with negative numbers for negative/unpleasant experiences and positive numbers for positive/pleasant experiences.
Evaluation of the level of psychological development | In the first interview, PTGI was applied to all pregnant women in all three groups as a pre-test at any time of pregnancy.
  PTGI (Post Traumatic Growth Inventory) was applied to determine the psychological development level of the pregnant women. PTGI is a 21-item Likert-type scale developed to evaluate positive changes after trauma and is scored between 0 and 5.
  The lowest score that can be obtained from the scale is 0, and the highest score is 105. A high score indicates that the person has experienced a high level of growth after the traumatic experience.
Evaluation of the level of psychological development | Seven day after the first interview, PTGI was applied to all pregnant women in all three groups as a post-test.
  PTGI (Post Traumatic Growth Inventory) was applied to determine the psychological development level of the pregnant women. PTGI is a 21-item Likert-type scale developed to evaluate positive changes after trauma and is scored between 0 and 5.
  The lowest score that can be obtained from the scale is 0, and the highest score is 105. A high score indicates that the person has experienced a high level of growth after the traumatic experience.
Evaluation of the level of well-being | In the first interview, WHO-5 well-being ındex was applied to all pregnant women in all three groups as a pre-test at any time of pregnancy.
  WHO-5 Well-Being Index was applied to determine the pwell-being level of the pregnant women. In order to determine mental well-being, the scale, which consists of 5 questions in total, is of 6-point Likert type, varying between "never", "sometimes", "less than half of the time", "more than half of the time" and "always". The raw score is calculated by adding the numbers of the five answers, and the resulting score ranges from zero to 25. Zero represents the worst possible quality of life and 25 the best possible quality of life.
Evaluation of the level of well-being | Seven day after the first interview, WHO-5 Well-Being IndexI was applied to all pregnant women in all three groups as a post-test.
  WHO-5 Well-Being Index was applied to determine the pwell-being level of the pregnant women. In order to determine mental well-being, the scale, which consists of 5 questions in total, is of 6-point Likert type, varying between "never", "sometimes", "less than half of the time", "more than half of the time" and "always". The raw score is calculated by adding the numbers of the five answers, and the resulting score ranges from zero to 25. Zero represents the worst possible quality of life and 25 the best possible quality of life.
Evaluation of the level of cortisol | At the first interview, saliva samples were taken from all pregnant women in all three groups as a pre-test at any time of pregnancy.
  Saliva samples were taken from pregnant women to determine the cortisol level. Saliva sample collection materials consist of 1.5 ml saliva collection tube (ependorf tube) and sips to facilitate the salivation process. The pregnant women were informed about the procedure to be followed and the saliva collection process was explained by the researcher.
  For salivary cortisol analysis, 96-well microplates were covered with cortisol-BSA at +4 C overnight and blocked with 200 µl BSA (1%) at 37 °C for 2 hours. Saliva samples were thawed before adding to microplates and centrifuged at 4000g for 10 minutes. The plates were incubated for 45 minutes at 37 °C and washed 5 times with washing solution. When the blue color occurred, the plates were read by the plate-reader spectrophotometer. Calibration curves were created using 4-parameter logistic regression curves and cortisol levels were measured using this curve.
Evaluation of the level of cortisol | Seven day after the first interview, saliva samples were taken from all pregnant women in all three groups as a post-test.
  Saliva samples were taken from pregnant women to determine the cortisol level. Saliva sample collection materials consist of 1.5 ml saliva collection tube (ependorf tube) and sips to facilitate the salivation process. The pregnant women were informed about the procedure to be followed and the saliva collection process was explained by the researcher.
  For salivary cortisol analysis, 96-well microplates were covered with cortisol-BSA at +4 C overnight and blocked with 200 µl BSA (1%) at 37 °C for 2 hours. Saliva samples were thawed before adding to microplates and centrifuged at 4000g for 10 minutes. The plates were incubated for 45 minutes at 37 °C and washed 5 times with washing solution. When the blue color occurred, the plates were read by the plate-reader spectrophotometer. Calibration curves were created using 4-parameter logistic regression curves and cortisol levels were measured using this curve.

CONTACTS AND LOCATIONS:
Overall Officials: Esra Karataş Okyay, Phd, Principal Investigator — Kahramanmaras Sutcu Imam University
Locations (1):
- Kahramanmaras Sutcu Imam University, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
we don't share individual participant data with other researchers

REFERENCES:
- [Result] Irmak Vural P, Aslan E. Emotional freedom techniques and breathing awareness to reduce childbirth fear: A randomized controlled study. Complement Ther Clin Pract. 2019 May;35:224-231. doi: 10.1016/j.ctcp.2019.02.011. Epub 2019 Feb 15. PMID 31003663
- See also: Description citation link — https://pubmed.ncbi.nlm.nih.gov/31003663/